CLINICAL TRIAL: NCT06940687
Title: Neurophysiological Benefits of Live Music for Early Alzheimer's Patients and Their Caregivers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Renée Fleming Foundation (Unknown); Yale University School of Medicine, Department of Psychiatry (Unknown); Howard University (Other); NeuroArts Blueprint Initiative (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000038702
Record Dates: First submitted 2025-02-19; First posted 2025-04-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease; Dementia; Mild Cognitive Impairment; Peer-bonded Caregiver; Caregiver
Keywords: Live Music; EEG; EKG/ECG; Anxiety; Connectedness; Social Connection
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Investigators aim to enroll 30 early Alzheimer's (AD) / Dementia / Mild Cognitive Impairment (MCI) participants and their 30 caregivers (30 dyads). A target sample size of 60 participants is proposed with an upper limit of 120 participants enrolled to allow for the possibility of losing a portion of the sample to follow-up.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AD / Dementia / MCI participants and caregivers dyads with music (Experimental): Each participant will take part in two sessions. Both sessions will last up to 3 hours.
  Participants will attend a series of live music performances and pre-recorded control session performances. Physiological and survey data will be collected to assess the impact of live versus pre-recorded music on anxiety, social motivation, parasympathetic activity, and neural synchrony.
  Interventions: Behavioral: Pre-recorded Music Session; Behavioral: Live Music Session

INTERVENTIONS:
Behavioral: Pre-recorded Music Session — A pre-recorded concert session
Behavioral: Live Music Session — A 45-minute live music performance

SUMMARY:
This study aims to investigate the neurophysiological effects of live music on individuals with early Alzheimer's Disease (AD), dementia, and/or mild cognitive impairment (MCI) and their caregivers. Heart rate (HR), heart rate variability (HRV), and brain activity will be measured as participant-caregiver dyads listen to preferred and improvised music performed by professional musicians. Investigators will leverage various measurement techniques including, but not limited to, electroencephalography (EEG), behavioral, surveys, and physiological monitoring to study the impact of live music on anxiety in AD and inter-dyad synchrony.

DETAILED DESCRIPTION:
Analysis of recordings captured during live concerts will be conducted using music information retrieval, pulse clarity, psychological ethnography, and similar methods. Investigators hypothesize that live music will reduce anxiety, increase social motivation, elevate parasympathetic activity, and enhance neural synchrony yielding increased interpersonal coordination, harmony, and emotional connection within dyads, indicating a positive impact on their autonomic nervous system and emotional well-being.

The primary objective of this study is to investigate the neurophysiological effects of live music concert experiences on people living with early AD and their caregivers using EEG and HR monitoring.

The secondary objectives of this study are to:

* Understand whether the live concert experience reduces state anxiety and enhances connection between individuals with early AD and their caregivers.
* Determine what role the physical characteristics of the concert music have on the wellbeing, behavior, connectedness, and autonomic function of people with early AD and their caregivers.

In-person sessions of the study will be conducted at a music / event venue in either the Greater New Haven, CT area, with possible expansion to venue(s) in the Washington, DC area, and/or the Nashville, TN area. The Yale IRB-approved study team may conduct the study at additional locations (including in the Washington, DC area and the Nashville, TN area) with permission from the venue(s).

Each participant will take part in two sessions. Both sessions will last up to 3 hours.

Participants will attend a series of live music performances and pre-recorded control session performances. Physiological and survey data will be collected to assess the impact of live versus pre-recorded music on anxiety, social motivation, parasympathetic activity, and neural synchrony.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Dementia Rating 0.5 - 2
* Be a person with or caregiver to a person with a diagnosis of early Alzheimer's Disease, mild dementia, and/or mild cognitive impairment (MCI)
* Able to provide informed consent
* Willing to wear an EEG headset and heart rate monitoring devices
* Willing to possibly have small patches of body / facial hair shaved to accommodate administration of heart rate monitoring devices
* Willing to answer survey questions about topics related to the study
* Willing to be audio / video recorded

Exclusion Criteria:

* Clinical Dementia Rating <0.5 or > 2
* Unable to provide informed consent
* Endorsing suicidal ideation (SI), self-injurious behavior, or homicidal ideation (HI) above the threshold defined in the "Risk Reduction and Safety Plan"
* Participating in another clinical trial studying AD and/or Dementia
* Starting a new prescription medication in the last 6 months
* Prescribed Benzodiazepines on an as needed basis

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2026-03-22 (Estimated); Study Completion 2026-03-22 (Estimated)

PRIMARY OUTCOMES:
Change in EEG activity during live music vs pre-recorded music conditions | Day 1 and Day 2, an average of 1 week apart
  EEG gamma measured by the Post Spectral Density measures in the gamma range (>30Hz) and theta (4-8Hz) frequency ranges during live music vs pre-recorded music conditions
motion capture | Day 1 and Day 2, an average of 1 week apart
  Capturing motion allows the researchers to investigate if patterns of bodily and stylistic characteristics of motion are associated with different emotional states in participants with Dementia and their caregivers. We will thematically analyze motion characteristics of and between individual participants during and between live and recorded music experiences using Laban Movement Analysis.
facial action units | Day 1 and Day 2, an average of 1 week apart
  Capturing facial expressions (i.e. facial action units) allows the researchers to study behavioral differences in emotion and arousal of and between individual participants exhibited during and between live and recorded music experiences.
eye gaze | Day 1 and Day 2, an average of 1 week apart
  Capturing eye gaze allows the researchers to study behavioral differences in attention and arousal of and between individual participants exhibited during and between live and recorded music experiences.
Changes in Standard Deviation of Normal-to-Normal (SDNN) Interval via electrocardiography (ECG, EKG). | Day 1 and Day 2, an average of 1 week apart
  Acquiring heart rate variability data via electrocardiography (ECG, EKG) allows the researchers to measure the standard deviation of Normal-to-Normal (SDNN) Interval in people with dementia, mild cognitive impairment, and/or Alzheimer's disease. SDNN Intervals measure both sympathetic and parasympathetic nervous system (SNS & PNS) responses (primarily sympathetic) in milliseconds.
Changes in Root Mean Square of Successive Differences (RMSSD) via electrocardiography (ECG, EKG). | Day 1 and Day 2, an average of 1 week apart
  Acquiring heart rate variability data via electrocardiography (ECG, EKG) allows the researchers to measure the Root Mean Square of Successive Differences (RMSSD) in people with dementia, mild cognitive impairment, and/or Alzheimer's disease. RMSSD measure parasympathetic responses in milliseconds.
Changes in Very low frequency (VLF) via electrocardiography (ECG, EKG). | Day 1 and Day 2, an average of 1 week apart
  Acquiring heart rate variability data via electrocardiography (ECG, EKG) allows the researchers to measure Very low frequency (VLF) in people with dementia, mild cognitive impairment, and/or Alzheimer's disease. VLF measure sympathetic responses in milliseconds squared.
Changes in the ratio of low frequency and high frequency (LF/HF) via electrocardiography (ECG, EKG). | Day 1 and Day 2, an average of 1 week apart
  Acquiring heart rate variability data via electrocardiography (ECG, EKG) allows the researchers to measure the ratio of low frequency (sympathetic response) and high frequency (parasympathetic response). This unitless measure is abbreviated as LF/HF and informs the researchers about the relationship between the SNS and PNS.

SECONDARY OUTCOMES:
music information retrieval (MIR) methods | Day 1 and Day 2, an average of 1 week apart
  Analyzing the physical characteristics of the music played during the sessions via music information retrieval (MIR) methods help the researchers make inferences about what music is effective in modulating wellbeing, connectedness, and behavior in this population.
Change in social connection using State Motivation to Foster Social Connections (SMFSCS)Scale | Day 1 and Day 2, an average of 1 week apart
  SMFSCS is a self-report questionnaire that measures the motivation individuals feel to form new connections and foster existing connection with others. 10 items on a 7-point Likert scale, from 1 (strongly disagree) to 7 (strongly agree). Total score is achieved by summing all items with total score range from 10-100. Higher scores indicate a greater motivation to create new connections and foster existing connections with others.
Change in absorption in music using the Absorption in Music Scale (AIMS) | Day 1 and Day 2, an average of 1 week apart
  SMFSCS is a self-report questionnaire that measures an individual's tendency to have strong emotional responses to music. 35 items on a 5-point Likert scale, from 1 (strongly disagree) to 5 (strongly agree). Total score is achieved by summing all items with total score range from 35-175. Higher scores indicate a greater tendency to have strong emotional responses to music.
Change in absorption in music using the Geriatric Anxiety Scale (GAS) | Day 1 and Day 2, an average of 1 week apart
  GAS is a self-report questionnaire that serves as a measure of anxiety for use with older adults. 30 items on a 5-point Likert scale, from 0 (not at all) to 3 (all of the time). Total score is achieved by summing items 1-25 with total score range from 0-75. Items 26 through 30 are used to help clinicians identify areas of concern for the respondent. Higher scores indicate more feelings of anxiety or stress.
Change in absorption in music using the State-Trait Anxiety Inventory (STAI) | Day 1 and Day 2, an average of 1 week apart
  STAI is a self-report questionnaire that measures transient and enduring levels of anxiety. 20 items on a 5-point Likert scale, from 1 (not at all) to 4 (very much so). Ten items are formed to record the presence of anxiety symptoms and the other 10 items are scored to record the absence of anxiety symptoms. Total score is achieved by summing all presence of anxiety items and inverting the absence of anxiety items with total score range from 20-80. Higher scores indicate higher levels transient and enduring anxiety.
Change in absorption in music using the Patient Health Questionnaire-9 (PHQ-9) | Day 1 and Day 2, an average of 1 week apart
  PHQ-9 is a self-report questionnaire that assesses 8 DSM-IV diagnoses, divided into threshold disorders and subthreshold disorders. 9 items on a 4-point Likert scale, from 0 (not at all) to 3 (nearly everyday). An item was also added to the end of the diagnostic portion of the PHQ-9 asking patients who checked off any problems on the questionnaire how difficult these symptoms make the respondent's life. Total score is achieved by summing all items with total score range from 0-27. Higher scores indicate higher depression severity.
Change in absorption in music using the Zarit Burden Interview (ZBI) | Day 1 and Day 2, an average of 1 week apart
  ZBI is a self-report questionnaire that measures the level of burden experienced by caregivers of patients with dementia. 22 items on a 5-point Likert scale, from 0 (never) to 4 (nearly always). Total score is achieved by summing all items with total score range from 0-88. Higher scores indicate greater burden.
Change in absorption in music using the Quality of Life Scale (QOLS) | Day 1 and Day 2, an average of 1 week apart
  QOLS is a self-report questionnaire that measures 5 conceptual domains of quality of life: material and physical well-being, relationships with other people, social, community and civic activities, personal development and fulfillment, and recreation. 16 items on a 7-point Likert scale, from 1 (terrible) to 7 (delighted). Total score is achieved by summing all items with total score range from 16-112. Higher scores indicate a greater satisfaction with life.

CONTACTS AND LOCATIONS:
Overall Officials: AZA Allsop, MD, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Firehouse 12 Studios, New Haven, Connecticut
  - Musical Intervention Studios, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No